CLINICAL TRIAL: NCT01475604
Title: Impact of Noninvasive Targeted Pulsed Electromagnetic Field (tPEMF) on Opioid Use, Pain, and Joint Function Following Total Knee Arthroplasty: A Double-Blind, Randomized, Sham-controlled Trial
Brief Title: Impact of Noninvasive Targeted Pulsed Electromagnetic Field (tPEMF) on Opioid Use, Pain, and Joint Function Following Total Knee Arthroplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Amp Orthopedics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IOH-TKA-001
Record Dates: First submitted 2011-11-17; First posted 2011-11-21 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Pulsed Radio Frequency, Electromagnetic Field therapy
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Magnetic Field Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Targeted pulsed electromagnetic field (Active Comparator)
  Interventions: Device: Ivivi Torino II
- Sham (Sham Comparator)
  Interventions: Device: Ivivi Torino II

INTERVENTIONS:
Device: Ivivi Torino II — Targeted pulsed electromagnetic field treatment for 4 weeks post-surgery
  Other Names: Electromagnetic Field Therapy
  Arms: Targeted pulsed electromagnetic field
Device: Ivivi Torino II — Sham treatment for 4 weeks post-surgery
  Other Names: Electromagnetic Field Therapy
  Arms: Sham

SUMMARY:
The purpose of this study is to determine the effectiveness of pulsed radio frequency (PRF), a type of electromagnetic field treatment with the Ivivi Torino II for reducing post-operative narcotic use in patients recovering from Total Knee Arthroplasty.

DETAILED DESCRIPTION:
Surgeons are continually looking for means to minimize postoperative pain following TKA in order to reduce or eliminate the need for opioid pain medications. Reductions in pain and edema along with improvements in range of motion encourage quicker recovery of joint function and normal activities. Pulsed radio frequency (PRF), a type of electromagnetic field treatment is proven to effectively modulate postoperative pain and edema in plastic surgery. Therefore, PRF has potential as an adjunct therapy for patients recovering from TKA.

The purpose of the current double-blind, randomized, sham-controlled clinical trial is to determine the effectiveness and safety of the Ivivi Torino II, a device that delivers pulsed radio frequency (PRF), a type of electromagnetic field treatment, in patients recovering from TKA for treatment of severe knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 80 years
* Primary diagnosis of knee OA
* Appropriate candidate for TKA
* Ability of the participant to comprehend the full nature and purpose of the study including possible risks and side effects
* Consent to the study and willing to comply with study product and methods including follow-up

Exclusion Criteria:

* Body mass index > 40 kg/m2
* Scheduled for bilateral TKA
* Advanced hip, spine, or ankle osteoarthritis that significantly limits ambulation
* Subjects who have any implanted metallic leads, wires, or systems (e.g. pacemaker, implantable cardioverter-defibrillator)
* Use of narcotic pain medication for any condition in the last 1 month prior to surgery
* Self-reported diagnosis of post-traumatic or inflammatory arthritis (e.g. rheumatoid or psoriatic)
* Pregnant or lactating female
* Participation in any clinical trial in the past 30 days
* Vulnerable populations including prisoners and nursing home residents
* Any medical condition that, in the opinion of the investigator, may compromise patient safety or confound the assessment of treatment effectiveness

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The average daily morphine equivalent dose consumption at 2 weeks post-surgery. | 2-week follow-up period from surgery

SECONDARY OUTCOMES:
Post-surgical opioid use during hospitalization and following discharge at 1 and 4 weeks post-surgery. | 1 and 4 weeks post-surgery
Knee pain severity assessed on a 10 cm visual analogue scale (VAS) | At intervals over the 4-week follow-up period
  Knee pain will be assessed for "current", pain at the time of data collection and "maximum", maximum pain experience at any point during the day of evaluation
The measurement of knee joint circumference | Measurement performed preoperatively, on the first or second postoperative day, at the discharge dressing change, and at the 4 week follow-up visit
  With patient in supine position, the circumference of the extended knee will be measured 1 cm proximal to the base of the patella using the same type of tape measure in all patients
Range of motion of the knee joint, assessed using the knee flexion technique | Assessed preoperatively, on the first or second postoperative day, at the discharge dressing change (unless discharged within 2 days), and at the 4 week follow-up visit
  Range of motion will be assessed using the knee flexion technique, which allows the use of a goniometer with the trans-epicondylar axis of the knee joint as the fulcrum.
OA-related medication use including analgesics, anti-inflammatories, and other non-opioids | 4 weeks post-surgery
  Subjects will be required to track daily OA-related medication use including analgesics, anti-inflammatories, and other non-opioids using a daily diary.
Adverse Events collected and analyzed for confirmation of device safety | Randomization to 4 weeks post-surgery
  Subjects will be instructed by the research staff and in the instructions in the daily diary to contact the research staff and/or investigator with any adverse events (AEs). Adverse events will be recorded daily.

CONTACTS AND LOCATIONS:
Overall Officials: Gerard A. Engh, M.D., Principal Investigator — Anderson Orthopaedic Research Institute
Locations (1):
- Anderson Orthopaedic Research Institute, Alexandria, Virginia, United States